CLINICAL TRIAL: NCT02238067
Title: Survey on Anemia Therapy With ESAs Medication in Chronic Kidney Disease Patients Not on Dialysis
Brief Title: Survey on Anemia Therapy in Participants With Chronic Kidney Disease (CKD) Not on Dialysis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25473
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-02

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Chronic Renal Anemia Participants: Participants with CKD who are not on dialysis and treated with ESA according to the usual standard of care and best practice guidelines, will be interviewed by physician who will complete the satisfaction surveys on anemia treatment at baseline and at 6 months follow-up visit.
  Interventions: Drug: ESA; Other: Satisfaction Survey Questionnaire

INTERVENTIONS:
Drug: ESA — Participants will continue to receive their ESA treatment, as per physician's discretion. The study protocol does not specify any particular ESA drug.
Other: Satisfaction Survey Questionnaire — Each participant will be interviewed to complete treatment satisfaction questionnaire survey at baseline and at 6-month follow-up visit.

SUMMARY:
This study is a prospective, non-interventional, cross-sectional multicenter survey. The aim is to better understand the current therapy pattern for anemia in CKD treated with erythropoiesis-stimulating agents (ESAs) and not on-dialysis participant population in Israel. Participating physicians will be requested to interview eligible participants with CKD not on dialysis and to complete for them a satisfaction survey for anemia treatment. The survey will be completed twice, once at study start and once at six months' follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants with CKD Stage 3-5
* Treated with ESAs
* Participant is speaking the same language as the investigator interviewer

Exclusion Criteria:

* Past or current treatment with dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with CKD not on-dialysis treated with ESAs
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2011-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- Israel (7):
  - Clalit- New Savyon Clinic, Ganey Tikva
  - Clalit - Diabetic HaMoshava South Clinic, Jerusalem
  - Clalit Carmiel, Karmiel
  - Clalit - Professional Clinic, Zvulun, Kiryat Bialik
  - Clalit Ben-Gurion, Naẕerat ‘Illit
  - Kaplan Medical Center; Nephrology and Hypertension Services, Rehovot
  - Clalit- Migdal HaMea Clinic, Tel Aviv, Tel Aviv

RESULTS

PARTICIPANT FLOW:
Groups:
- Chronic Renal Anemia Participants: Participants with Chronic Kidney Disease (CKD) who were not on dialysis and treated with Erythropoiesis-Stimulating Agents (ESA) according to the usual standard of care and best practice guidelines, were interviewed by physician who completed the satisfaction surveys on anemia treatment at baseline and at 6 months follow-up visit.
Period: Overall Study
Arm/Group | Chronic Renal Anemia Participants
Started | 196
Completed | 151
Not Completed | 45
Not completed — Not completed survey at Month 6 | 45

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Chronic Renal Anemia Participants: Participants with CKD who were not on dialysis and treated with ESA according to the usual standard of care and best practice guidelines, were interviewed by physician who completed the satisfaction surveys on anemia treatment at baseline and at 6 months follow-up visit.
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 196
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.6 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 111

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants by ESA Types at Baseline
Description: Assessment was performed by physician via a satisfaction survey on anemia treatment. ESA types included: Mircera, Recormon, Eprex, and Aranesp. Percentage of participants with each ESA type was reported.
Time Frame: Baseline
Population: All enrolled participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 196
percentage of participants
  Mircera | 51.5 [44.3 to 58.7]
  Recormon | 17.3 [12.3 to 23.4]
  Eprex | 10.7 [6.8 to 15.9]
  Aranesp | 20.4 [15.0 to 26.7]

2. Primary Outcome: Percentage of Participants by ESA Types at Month 6
Description: as for outcome 1
Time Frame: Month 6
Population: All enrolled participants who completed the questionnaire at Month 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 151
percentage of participants
  Mircera | 43.7 [35.7 to 52.0]
  Recormon | 19.2 [13.3 to 26.4]
  Eprex | 12.6 [7.7 to 19.0]
  Aranesp | 24.5 [17.9 to 32.2]

3. Primary Outcome: Percentage of Participants by Frequency of ESA Use at Baseline
Description: Assessment was performed by physician via a satisfaction survey on anemia treatment. Frequency of ESA use included:Three times a week, twice a week, once a week, every 2 weeks, every 4 weeks or other (any other frequency). Percentage of participants by each frequency of ESA use was reported.
Time Frame: Baseline
Population: All enrolled participants. Number of participants analyzed = participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 195
percentage of participants
  Three times a week | 2.6 [0.8 to 5.9]
  Twice a week | 7.2 [4.0 to 11.8]
  Once a week | 14.9 [10.2 to 20.7]
  Every 2 weeks | 26.2 [20.1 to 32.9]
  Every 4 weeks | 38.5 [31.6 to 45.7]
  Other | 10.8 [6.8 to 16.0]

4. Primary Outcome: Percentage of Participants by Frequency of ESA Use at Month 6
Description: as for outcome 3
Time Frame: Month 6
Population: All enrolled participants who completed the questionnaire at Month 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 151
percentage of participants
  Three times a week | 1.3 [0.2 to 4.7]
  Twice a week | 4.0 [1.5 to 8.4]
  Once a week | 15.9 [10.5 to 22.7]
  Every 2 weeks | 25.2 [18.5 to 32.9]
  Every 4 weeks | 39.1 [31.2 to 47.3]
  Other | 14.6 [9.4 to 21.2]

5. Primary Outcome: Percentage of Participants by Frequency and Types of ESA Used at Baseline
Description: Assessment was performed by physician via a satisfaction survey on anemia treatment. Frequency of ESA use included:Three times a week, twice a week, once a week, every 2 weeks, every 4 weeks or other (any other frequency). ESA types included: Mircera, Recormon, Eprex, and Aranesp. Percentage of participants with each ESA type and each frequency of ESA use was reported.
Time Frame: Baseline
Population: All enrolled participants. Number of participants analyzed = participants evaluable for this outcome measure. Here 'n' signifies number of participants evaluable for specified categories.
Measure: Number; unit: percentage of participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 195
percentage of participants
  Mircera : Three times a week (n=100) | 2.0
  Mircera : Twice a week (n=100) | 4.0
  Mircera : Once a week (n=100) | 1.0
  Mircera : Every 2 weeks (n=100) | 26.0
  Mircera : Every 4 weeks (n=100) | 67.0
  Mircera : Other (n=100) | 0
  Recormon : Three times a week (n=34) | 0
  Recormon : Twice a week (n=34) | 17.6
  Recormon : Once a week (n=34) | 38.2
  Recormon : Every 2 weeks (n=34) | 17.6
  Recormon : Every 4 weeks (n=34) | 5.9
  Recormon : Other (n=34) | 20.6
  Eprex : Three times a week (n=21) | 9.5
  Eprex : Twice a week (n=21) | 9.5
  Eprex : Once a week (n=21) | 42.9
  Eprex : Every 2 weeks (n=21) | 9.5
  Eprex : Every 4 weeks (n=21) | 4.8
  Eprex : Other (n=21) | 23.8
  Aranesp : Three times a week (n=40) | 2.5
  Aranesp : Twice a week (n=40) | 5.0
  Aranesp : Once a week (n=40) | 15.0
  Aranesp : Every 2 weeks (n=40) | 42.5
  Aranesp : Every 4 weeks (n=40) | 12.5
  Aranesp : Other (n=40) | 22.5

6. Primary Outcome: Percentage of Participants by Frequency and Types of ESA Used at Month 6
Description: as for outcome 5
Time Frame: Month 6
Population: All enrolled participants who completed the questionnaire at Month 6. Here 'n' signifies number of participants evaluable for specified categories.
Measure: Number; unit: percentage of participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 151
percentage of participants
  Mircera : Three times a week (n=66) | 1.5
  Mircera : Twice a week (n=66) | 1.5
  Mircera : Once a week (n=66) | 0
  Mircera : Every 2 weeks (n=66) | 18.2
  Mircera : Every 4 weeks (n=66) | 71.2
  Mircera : Other (n=66) | 7.6
  Recormon : Three times a week (n=29) | 0
  Recormon : Twice a week (n=29) | 10.3
  Recormon : Once a week (n=29) | 27.6
  Recormon : Every 2 weeks (n=29) | 37.9
  Recormon : Every 4 weeks (n=29) | 6.9
  Recormon : Other (n=29) | 17.2
  Eprex : Three times a week (n=19) | 5.3
  Eprex : Twice a week (n=19) | 5.3
  Eprex : Once a week (n=19) | 47.4
  Eprex : Every 2 weeks (n=19) | 15.8
  Eprex : Every 4 weeks (n=19) | 5.3
  Eprex : Other (n=19) | 21.1
  Aranesp : Three times a week (n=37) | 0
  Aranesp : Twice a week (n=37) | 2.7
  Aranesp : Once a week (n=37) | 18.9
  Aranesp : Every 2 weeks (n=37) | 32.4
  Aranesp : Every 4 weeks (n=37) | 24.3
  Aranesp : Other (n=37) | 21.6

7. Secondary Outcome: Percentage of Participants by Different CKD Stages
Description: Assessment was performed by physician via a satisfaction survey on anemia treatment. CKD stages were based on participant's answer to the survey question. No specific method of assessment for CKD stage was specified. Percentage of participants with each CKD stage was reported.
Time Frame: Baseline, Month 6
Population: All enrolled participants. Here 'n' signifies number of participants evaluable at specified time-points.
Measure: Number; unit: percentage of participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 196
percentage of participants
  Stage 1 : Baseline (n=196) | 2.0
  Stage 1 : Month 6 (n=151) | 1.3
  Stage 2 : Baseline (n=196) | 10.2
  Stage 2 : Month 6 (n=151) | 13.9
  Stage 3 : Baseline (n=196) | 37.8
  Stage 3 : Month 6 (n=151) | 41.7
  Stage 4 : Baseline (n=196) | 37.8
  Stage 4 : Month 6 (n=151) | 30.5
  Stage 5 : Baseline (n=196) | 12.2
  Stage 5 : Month 6 (n=151) | 12.6

8. Secondary Outcome: Percentage of Participants by Different Injection Administration Modes
Description: Assessment was performed by physician via a satisfaction survey on anemia treatment. Participants were asked: 'How do you currently inject the anemia treatment?' and reported any of the 5 possible answers: Independently, by a family member, nurse at home, nurse at the clinic or other. Percentage of participants with each injection administration modes was reported.
Time Frame: Baseline, Month 6
Population: All enrolled participants. Here 'n' signifies number of participants evaluable at specified time-points.
Measure: Number; unit: percentage of participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 196
percentage of participants
  Independently : Baseline (n=196) | 18.4
  Independently : Month 6 (n=151) | 23.2
  By a family member : Baseline (n=196) | 16.8
  By a family member : Month 6 (n=151) | 17.9
  Nurse at home : Baseline (n=196) | 3.6
  Nurse at home : Month 6 (n=151) | 3.3
  Nurse at the clinic : Baseline (n=196) | 58.2
  Nurse at the clinic : Month 6 (n=151) | 52.3
  Other: Baseline (n=196) | 3.1
  Other : Month 6 (n=151) | 3.3

9. Secondary Outcome: Percentage of Participants With Interest in Learning to Inject Independently
Description: Assessment was performed by physician via a satisfaction survey on anemia treatment. Participants responded 'yes' or 'no' to the question: 'Would you be interested in learning to inject independently?' ' Percentage of participants who responded 'yes', was reported.
Time Frame: Baseline, Month 6
Population: All enrolled participants who did not inject independently. Here 'n' signifies number of participants evaluable at specified time-points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 160
percentage of participants
  Baseline (n=160) | 6.3 [3.0 to 11.2]
  Month 6 (n=116) | 4.3 [1.4 to 9.8]

10. Secondary Outcome: Percentage of Participants by Need for Improvement in Treatment Frequency
Description: Assessment was performed by physician via a satisfaction survey on anemia treatment. Participants were asked to rate their need for improvement in the frequency of treatment received currently on a 1-5 scale, where 1 represents 'Convenient, there is no need for improvement' and 5 represents 'Improvement is very necessary'. Percentage of participants with each score was reported.
Time Frame: Baseline, Month 6
Population: All enrolled participants. Here 'n' signifies number of participants evaluable at specified time-points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 196
percentage of participants
  Score 1 : Baseline (n=196) | 94.9 [90.8 to 97.5]
  Score 1 : Month 6 (n=151) | 96.0 [91.6 to 98.5]
  Score 2 : Baseline (n=196) | 1.5 [0.3 to 4.4]
  Score 2 : Month 6 (n=151) | 1.3 [0.2 to 4.7]
  Score 3 : Baseline (n=196) | 1.5 [0.3 to 4.4]
  Score 3 : Month 6 (n=151) | 1.3 [0.2 to 4.7]
  Score 4 : Baseline (n=196) | 1.5 [0.3 to 4.4]
  Score 4 : Month 6 (n=151) | 0.7 [0 to 3.6]
  Score 5 : Baseline (n=196) | 0.5 [0 to 2.8]
  Score 5 : Month 6 (n=151) | 0.7 [0 to 3.6]

11. Secondary Outcome: Percentage of Participants by Need for Improvement in Treatment Frequency by ESA Type
Description: Assessment was performed by physician via a satisfaction survey on anemia treatment. Participants were asked for the type of ESA received (Mircera, Recormon, Eprex or Aranesp) and to rate their need for improvement in the frequency of each treatment received currently on a 1-5 scale, where 1 represents 'Convenient, there is no need for improvement' and 5 represents 'improvement is very necessary'. Percentage of participants with each score and ESA type was reported.
Time Frame: Baseline, Month 6
Population: All enrolled participants. Here 'n' signifies number of participants evaluable for specified categories.
Measure: Number; unit: percentage of participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 196
percentage of participants
  Mircera: Score 1: Baseline (n=101) | 98.0
  Mircera: Score 2: Baseline (n=101) | 2.0
  Mircera: Score 3: Baseline (n=101) | 0
  Mircera: Score 4: Baseline (n=101) | 0
  Mircera: Score 5: Baseline (n=101) | 0
  Recormon: Score 1: Baseline (n=34) | 94.1
  Recormon: Score 2: Baseline (n=34) | 0
  Recormon: Score 3: Baseline (n=34) | 0
  Recormon: Score 4: Baseline (n=34) | 2.9
  Recormon: Score 5: Baseline (n=34) | 2.9
  Eprex: Score 1: Baseline (n=21) | 90.5
  Eprex: Score 2: Baseline (n=21) | 0
  Eprex: Score 3: Baseline (n=21) | 9.5
  Eprex: Score 4: Baseline (n=21) | 0
  Eprex: Score 5: Baseline (n=21) | 0
  Aranesp: Score 1: Baseline (n=40) | 90.0
  Aranesp: Score 2: Baseline (n=40) | 2.5
  Aranesp: Score 3: Baseline (n=40) | 2.5
  Aranesp: Score 4: Baseline (n=40) | 5.0
  Aranesp: Score 5: Baseline (n=40) | 0
  Mircera: Score 1: Month 6 (n=66) | 100.0
  Mircera: Score 2: Month 6 (n=66) | 0
  Mircera: Score 3: Month 6 (n=66) | 0
  Mircera: Score 4: Month 6 (n=66) | 0
  Mircera: Score 5: Month 6 (n=66) | 0
  Recormon: Score 1: Month 6 (n=29) | 96.6
  Recormon: Score 2: Month 6 (n=29) | 0
  Recormon: Score 3: Month 6 (n=29) | 3.4
  Recormon: Score 4: Month 6 (n=29) | 0
  Recormon: Score 5: Month 6 (n=29) | 0
  Eprex: Score 1: Month 6 (n=19) | 94.7
  Eprex: Score 2: Month 6 (n=19) | 5.3
  Eprex: Score 3: Month 6 (n=19) | 0
  Eprex: Score 4: Month 6 (n=19) | 0
  Eprex: Score 5: Month 6 (n=19) | 0
  Aranesp: Score 1: Month 6 (n=37) | 89.2
  Aranesp: Score 2: Month 6 (n=37) | 2.7
  Aranesp: Score 3: Month 6 (n=37) | 2.7
  Aranesp: Score 4: Month 6 (n=37) | 2.7
  Aranesp: Score 5: Month 6 (n=37) | 2.7

12. Secondary Outcome: Percentage of Participants by Preferred Treatment Frequency
Description: Assessment was performed by physician via a satisfaction survey on anemia treatment. Participants were asked "Assuming that there are several options for anemia treatment with the only difference being the frequency of use, what is your preference?". Participants answered as either once a month, twice a month, once a week, twice a week, three times a week or other (any other frequency). Percentage of participants with each preferred treatment frequency was reported.
Time Frame: Baseline, Month 6
Population: All enrolled participants. Here 'n' signifies number of participants evaluable at specified time-points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 196
percentage of participants
  Once a month: Baseline (n=196) | 63.8 [56.6 to 70.5]
  Once a month: Month 6 (n=151) | 49.0 [40.8 to 57.3]
  Twice a month: Baseline (n=196) | 17.3 [12.3 to 23.4]
  Twice a month: Month 6 (n=151) | 23.8 [17.3 to 31.4]
  Once a week: Baseline (n=196) | 12.8 [8.4 to 18.3]
  Once a week: Month 6 (n=151) | 17.2 [11.6 to 24.2]
  Twice a week: Baseline (n=196) | 2.0 [0.6 to 5.1]
  Twice a week: Month 6 (n=151) | 2.0 [0.4 to 5.7]
  Three times a week: Baseline (n=196) | 1.0 [0.1 to 3.6]
  Three times a week: Month 6 (n=151) | 0.7 [0 to 3.6]
  Other: Baseline (n=196) | 3.1 [1.1 to 6.5]
  Other: Month 6 (n=151) | 7.3 [3.7 to 12.7]

13. Secondary Outcome: Percentage of Participants by Preferred Treatment Frequency by ESA Type
Description: Assessment was performed by physician via a satisfaction survey on anemia treatment. Participants were asked for the type of ESA received (Mircera, Recormon, Eprex or Aranesp) and their preference of treatment frequency. Participants were asked "Assuming that there are several options for anemia treatment with the only difference being the frequency of use, what is your preference?". Participants answered as either once a month, twice a month, once a week, twice a week, three times a week or other (any other frequency). Percentage of participants with each preferred treatment frequency and ESA type was reported.
Time Frame: Baseline, Month 6
Population: All enrolled participants. Here 'n' signifies number of participants evaluable for specified categories.
Measure: Number; unit: percentage of participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 196
percentage of participants
  Mircera: Once a month: Baseline (n=101) | 83.2
  Mircera: Once a month: Month 6 (n=66) | 75.8
  Mircera: Twice a month: Baseline (n=101) | 14.9
  Mircera: Twice a month: Month 6 (n=66) | 15.2
  Mircera: Once a week: Baseline (n=101) | 1.0
  Mircera: Once a week: Month 6 (n=66) | 3.0
  Mircera: Twice a week: Baseline (n=101) | 1.0
  Mircera: Twice a week: Month 6 (n=66) | 0
  Mircera: Three times a week: Baseline (n=101) | 0
  Mircera: Three times a week: Month 6 (n=66) | 0
  Mircera: Other: Baseline (n=101) | 0
  Mircera: Other: Month 6 (n=66) | 6.1
  Recormon: Once a month: Baseline (n=34) | 44.1
  Recormon: Once a month: Month 6 (n=29) | 27.6
  Recormon: Twice a month: Baseline (n=34) | 14.7
  Recormon: Twice a month: Month 6 (n=29) | 31.0
  Recormon: Once a week: Baseline (n=34) | 35.3
  Recormon: Once a week: Month 6 (n=29) | 31.0
  Recormon: Twice a week: Baseline (n=34) | 2.9
  Recormon: Twice a week: Month 6 (n=29) | 6.9
  Recormon: Three times a week: Baseline (n=34) | 0
  Recormon: Three times a week: Month 6 (n=29) | 3.4
  Recormon: Other: Baseline (n=34) | 2.9
  Recormon: Other: Month 6 (n=29) | 0
  Eprex: Once a month: Baseline (n=21) | 33.3
  Eprex: Once a month: Month 6 (n=19) | 10.5
  Eprex: Twice a month: Baseline (n=21) | 0
  Eprex: Twice a month: Month 6 (n=19) | 15.8
  Eprex: Once a week: Baseline (n=21) | 42.9
  Eprex: Once a week: Month 6 (n=19) | 52.6
  Eprex: Twice a week: Baseline (n=21) | 9.5
  Eprex: Twice a week: Month 6 (n=19) | 5.3
  Eprex: Three times a week: Baseline (n=21) | 4.8
  Eprex: Three times a week: Month 6 (n=19) | 0
  Eprex: Other: Baseline (n=21) | 9.5
  Eprex: Other: Month 6 (n=19) | 15.8
  Aranesp: Once a month: Baseline (n=40) | 47.5
  Aranesp: Once a month: Month 6 (n=37) | 37.8
  Aranesp: Twice a month: Baseline (n=40) | 35.0
  Aranesp: Twice a month: Month 6 (n=37) | 37.8
  Aranesp: Once a week: Baseline (n=40) | 7.5
  Aranesp: Once a week: Month 6 (n=37) | 13.5
  Aranesp: Twice a week: Baseline (n=40) | 0
  Aranesp: Twice a week: Month 6 (n=37) | 0
  Aranesp: Three times a week: Baseline (n=40) | 2.5
  Aranesp: Three times a week: Month 6 (n=37) | 0
  Aranesp: Other: Baseline (n=40) | 7.5
  Aranesp: Other: Month 6 (n=37) | 10.8

14. Secondary Outcome: Percentage of Participants by Preferred Treatment Frequency by Baseline ESA Frequency
Description: Assessment was performed by physician via a satisfaction survey on anemia treatment. Participants were asked for their preference of treatment frequency and baseline ESA frequency. Participants were asked "Assuming that there are several options for anemia treatment with the only difference being the frequency of use, what is your preference?". Preferred treatment frequency included: once a month (O/M), twice a month (B/M), once a week (O/W), twice a week (B/W), three times a week (T/W) or other (any other frequency]). Frequency of baseline ESA use included: three times a week, twice a week, once a week, every 2 weeks (Q2W), every 4 weeks (Q4W) or other (any other frequency). Percentage of participants by each preferred treatment frequency and baseline ESA frequency was reported.
Time Frame: Baseline, Month 6
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 195
percentage of participants
  Preferred O/M: Baseline ESA T/W: Baseline (n=5) | 80.0
  Preferred O/M: Baseline ESA T/W: Month 6 (n=2) | 50.0
  Preferred O/M: Baseline ESA B/W: Baseline (n=14) | 28.6
  Preferred O/M: Baseline ESA B/W: Month 6 (n=6) | 0
  Preferred O/M: Baseline ESA O/W: Baseline (n=29) | 27.6
  Preferred O/M: Baseline ESA O/W: Month 6 (n=24) | 12.5
  Preferred O/M: Baseline ESA Q2W: Baseline (n=51) | 49.0
  Preferred O/M: Baseline ESA Q2W: Month 6 (n=38) | 13.2
  Preferred O/M: Baseline ESA Q4W: Baseline (n=75) | 98.7
  Preferred O/M: Baseline ESA Q4W: Month 6 (n=59) | 96.6
  Preferred O/M: Baseline ESA other: Baseline (n=21) | 47.6
  Preferred O/M: Baseline ESA other: Month 6 (n=22) | 36.4
  Preferred B/M: Baseline ESA T/W: Baseline (n=5) | 0
  Preferred B/M: Baseline ESA T/W: Month 6 (n=2) | 0
  Preferred B/M: Baseline ESA B/W: Baseline (n=14) | 28.6
  Preferred B/M: Baseline ESA B/W: Month 6 (n=6) | 33.3
  Preferred B/M: Baseline ESA O/W: Baseline (n=29) | 10.3
  Preferred B/M: Baseline ESA O/W: Month 6 (n=24) | 8.3
  Preferred B/M: Baseline ESA Q2W: Baseline (n=51) | 47.1
  Preferred B/M: Baseline ESA Q2W: Month 6 (n=38) | 81.6
  Preferred B/M: Baseline ESA Q4W: Baseline (n=75) | 0
  Preferred B/M: Baseline ESA Q4W: Month 6 (n=59) | 0
  Preferred B/M: Baseline ESA other: Baseline (n=21) | 9.5
  Preferred B/M: Baseline ESA other: Month 6 (n=22) | 4.5
  Preferred O/W: Baseline ESA T/W: Baseline (n=5) | 0
  Preferred O/W: Baseline ESA T/W: Month 6 (n=2) | 50.0
  Preferred O/W: Baseline ESA B/W: Baseline (n=14) | 28.6
  Preferred O/W: Baseline ESA B/W: Month 6 (n=6) | 33.3
  Preferred O/W: Baseline ESA O/W: Baseline (n=29) | 62.1
  Preferred O/W: Baseline ESA O/W: Month 6 (n=24) | 79.2
  Preferred O/W: Baseline ESA Q2W: Baseline (n=51) | 2.0
  Preferred O/W: Baseline ESA Q2W: Month 6 (n=38) | 2.6
  Preferred O/W: Baseline ESA Q4W: Baseline (n=75) | 0
  Preferred O/W: Baseline ESA Q4W: Month 6 (n=59) | 1.7
  Preferred O/W: Baseline ESA other: Baseline (n=21) | 9.5
  Preferred O/W: Baseline ESA other: Month 6 (n=22) | 9.1
  Preferred B/W: Baseline ESA T/W: Baseline (n=5) | 0
  Preferred B/W: Baseline ESA T/W: Month 6 (n=2) | 0
  Preferred B/W: Baseline ESA B/W: Baseline (n=14) | 14.3
  Preferred B/W: Baseline ESA B/W: Month 6 (n=6) | 33.3
  Preferred B/W: Baseline ESA O/W: Baseline (n=29) | 0
  Preferred B/W: Baseline ESA O/W: Month 6 (n=24) | 0
  Preferred B/W: Baseline ESA Q2W: Baseline (n=51) | 2.0
  Preferred B/W: Baseline ESA Q2W: Month 6 (n=38) | 2.6
  Preferred B/W: Baseline ESA Q4W: Baseline (n=75) | 0
  Preferred B/W: Baseline ESA Q4W: Month 6 (n=59) | 0
  Preferred B/W: ESA other: Baseline (n=21) | 4.8
  Preferred B/W: ESA other: Month 6 (n=22) | 0
  Preferred T/W: Baseline ESA T/W: Baseline (n=5) | 20.0
  Preferred T/W: Baseline ESA T/W: Month 6 (n=2) | 0
  Preferred T/W: Baseline ESA B/W: Baseline (n=14) | 0
  Preferred T/W: Baseline ESA B/W: Month 6 (n=6) | 0
  Preferred T/W: Baseline ESA O/W: Baseline (n=29) | 0
  Preferred T/W: Baseline ESA O/W: Month 6 (n=24) | 0
  Preferred T/W: Baseline ESA Q2W: Baseline (n=51) | 0
  Preferred T/W: Baseline ESA Q2W: Month 6 (n=38) | 0
  Preferred T/W: Baseline ESA Q4W: Baseline (n=75) | 1.3
  Preferred T/W: Baseline ESA Q4W: Month 6 (n=59) | 1.7
  Preferred T/W: Baseline ESA other: Baseline (n=21) | 0
  Preferred T/W: Baseline ESA other: Month 6 (n=22) | 0
  Preferred Other: Baseline ESA T/W: Baseline (n=5) | 0
  Preferred Other: Baseline ESA T/W: Month 6 (n=2) | 0
  Preferred Other: Baseline ESA B/W: Baseline (n=14) | 0
  Preferred Other: Baseline ESA B/W: Month 6 (n=6) | 0
  Preferred Other: Baseline ESA O/W: Month 6 (n=29) | 0
  Preferred Other: Baseline ESA O/W: Month 6 (n=24) | 0
  Preferred Other: Baseline ESA Q2W: Baseline (n=51) | 0
  Preferred Other: Baseline ESA Q2W: Month 6 (n=38) | 0
  Preferred Other: Baseline ESA Q4W: Baseline (n=75) | 0
  Preferred Other: Baseline ESA Q4W: Month 6 (n=59) | 0
  Preferred Other:Baseline ESA other:Baseline (n=21) | 28.6
  Preferred Other:Baseline ESA other: Month 6 (n=22) | 50.0

15. Secondary Outcome: Percentage of Participants by Limitation of Daily Life Due to ESA Refrigeration Requirements
Description: Assessment was performed by physician via a satisfaction survey on anemia treatment. Participants were asked to rate their limitation of daily life due to ESA refrigeration requirements on a 1-5 scale, where 1 represents 'Does not limit' and 5 represents 'significantly limits'. Percentage of participants with each score was reported.
Time Frame: Baseline, Month 6
Population: All enrolled participants. Here 'n' signifies number of participants evaluable at specified time-points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 196
percentage of participants
  Score 1: Baseline (n=196) | 96.4 [92.8 to 98.6]
  Score 1: Month 6 (n=151) | 97.4 [93.4 to 99.3]
  Score 2: Baseline (n=196) | 1.0 [0.1 to 3.6]
  Score 2: Month 6 (n=151) | 0.7 [0 to 3.6]
  Score 3: Baseline (n=196) | 0 [0 to 0]
  Score 3: Month 6 (n=151) | 1.3 [0.2 to 4.7]
  Score 4: Baseline (n=196) | 0.5 [0 to 2.8]
  Score 4: Month 6 (n=151) | 0 [0 to 0]
  Score 5: Baseline (n=196) | 2.0 [0.6 to 5.1]
  Score 5: Month 6 (n=151) | 0.7 [0 to 3.6]

16. Secondary Outcome: Percentage of Participants by Limitation of Daily Life Due to ESA Refrigeration Requirements by ESA Types
Description: Assessment was performed by physician via a satisfaction survey on anemia treatment. Participants were asked for the type of ESA received (Mircera, Recormon, Eprex or Aranesp) and to rate their limitation of daily life due to ESA refrigeration requirements on a 1-5 scale, where 1 represents 'Does not limit' and 5 represents 'significantly limits'. Percentage of participants with each score and ESA type was reported.
Time Frame: Baseline, Month 6
Population: All enrolled participants. Here 'n' signifies number of participants evaluable for specified categories.
Measure: Number; unit: percentage of participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 196
percentage of participants
  Mircera: Score 1: Baseline (n=101) | 97.0
  Mircera: Score 2: Baseline (n=101) | 1.0
  Mircera: Score 4: Baseline (n=101) | 0
  Mircera: Score 5: Baseline (n=101) | 2.0
  Mircera: Score 1: Month 6 (n=66) | 100.0
  Mircera: Score 2: Month 6 (n=66) | 0
  Mircera: Score 3: Month 6 (n=66) | 0
  Mircera: Score 5: Month 6 (n=66) | 0
  Recormon: Score 1: Baseline (n=34) | 100.0
  Recormon: Score 2: Baseline (n=34 | 0
  Recormon: Score 4: Baseline (n=34 | 0
  Recormon: Score 5: Baseline (n=34 | 0
  Recormon: Score 1: Month 6 (n=29) | 96.6
  Recormon: Score 2: Month 6 (n=29) | 3.4
  Recormon: Score 3: Month 6 (n=29) | 0
  Recormon: Score 5: Month 6 (n=29) | 0
  Eprex: Score 1: Baseline (n=21) | 100.0
  Eprex: Score 2: Baseline (n=21) | 0
  Eprex: Score 4: Baseline (n=21) | 0
  Eprex: Score 5: Baseline (n=21) | 0
  Eprex: Score 1: Month 6 (n=19) | 94.7
  Eprex: Score 2: Month 6 (n=19) | 0
  Eprex: Score 3: Month 6 (n=19) | 0
  Eprex: Score 5: Month 6 (n=19) | 5.3
  Aranesp: Score 1: Baseline (n=40) | 90.0
  Aranesp: Score 2: Baseline (n=40) | 2.5
  Aranesp: Score 4: Baseline (n=40) | 2.5
  Aranesp: Score 5: Baseline (n=40) | 5.0
  Aranesp: Score 1: Month 6 (n=37) | 94.6
  Aranesp: Score 2: Month 6 (n=37) | 0
  Aranesp: Score 3: Month 6 (n=37) | 5.4
  Aranesp: Score 5: Month 6 (n=37) | 0

17. Secondary Outcome: Percentage of Participants by Convenience of Syringe Usage
Description: Assessment was performed by physician via a satisfaction survey on anemia treatment. Participants were asked to rate their convenience of syringe usage on a 1-5 scale, where 1 represents 'Inconvenient' and 5 represents 'Very convenient'. Percentage of participants with each score was reported.
Time Frame: Baseline, Month 6
Population: All enrolled participants. Here 'n' signifies number of participants evaluable at specified time-points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 196
percentage of participants
  Score 1: Baseline (n=196) | 2.0 [0.6 to 5.1]
  Score 3: Baseline (n=196) | 2.6 [0.8 to 5.9]
  Score 4: Baseline (n=196) | 6.6 [3.6 to 11.1]
  Score 5: Baseline (n=196) | 88.8 [83.5 to 92.8]
  Score 1: Month 6 (n=151) | 0.7 [0 to 3.6]
  Score 3: Month 6 (n=151) | 2.0 [0.4 to 5.7]
  Score 4: Month 6 (n=151) | 4.0 [1.5 to 8.4]
  Score 5: Month 6 (n=151) | 93.4 [88.2 to 96.8]

18. Secondary Outcome: Percentage of Participants by Convenience of Syringe Usage by ESA Type
Description: Assessment was performed by physician via a satisfaction survey on anemia treatment. Participants were asked for the type of ESA received (Mircera, Recormon, Eprex or Aranesp) and to rate their convenience of syringe usage on a 1-5 scale, where 1 represents 'Inconvenient' and 5 represents 'Very convenient'. Percentage of participants with each score and ESA type was reported.
Time Frame: Baseline, Month 6
Population: All enrolled participants. Here 'n' signifies number of participants evaluable for specified categories.
Measure: Number; unit: percentage of participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 196
percentage of participants
  Mircera: Score 1: Baseline (n=101) | 4.0
  Mircera: Score 3: Baseline (n=101) | 1.0
  Mircera: Score 4: Baseline (n=101) | 5.0
  Mircera: Score 5: Baseline (n=101) | 90.1
  Mircera: Score 1: Month 6 (n=66) | 0
  Mircera: Score 3: Month 6 (n=66) | 0
  Mircera: Score 4: Month 6 (n=66) | 1.5
  Mircera: Score 5: Month 6 (n=66) | 98.5
  Recormon: Score 1: Baseline (n=34) | 0
  Recormon: Score 3: Baseline (n=34) | 2.9
  Recormon: Score 4: Baseline (n=34) | 11.8
  Recormon: Score 5: Baseline (n=34) | 85.3
  Recormon: Score 1: Month 6 (n=29) | 0
  Recormon: Score 3: Month 6 (n=29) | 3.4
  Recormon: Score 4: Month 6 (n=29) | 6.9
  Recormon: Score 5: Month 6 (n=29) | 89.7
  Eprex: Score 1: Baseline (n=21) | 0
  Eprex: Score 3: Baseline (n=21) | 0
  Eprex: Score 4: Baseline (n=21) | 0
  Eprex: Score 5: Baseline (n=21) | 100.0
  Eprex: Score 1: Month 6 (n=19) | 5.3
  Eprex: Score 3: Month 6 (n=19) | 5.3
  Eprex: Score 4: Month 6 (n=19) | 0
  Eprex: Score 5: Month 6 (n=19) | 89.5
  Aranesp: Score 1: Baseline (n=40) | 0
  Aranesp: Score 3: Baseline (n=40) | 7.5
  Aranesp: Score 4: Baseline (n=40) | 10.0
  Aranesp: Score 5: Baseline (n=40) | 82.5
  Aranesp: Score 1: Month 6 (n=37) | 0
  Aranesp: Score 3: Month 6 (n=37) | 2.7
  Aranesp: Score 4: Month 6 (n=37) | 8.1
  Aranesp: Score 5: Month 6 (n=37) | 89.2

19. Secondary Outcome: Percentage of Participants by Injection Site Pain
Description: Assessment was performed by physician via a satisfaction survey on anemia treatment. Participants were asked to rate their injection site pain on a 1-5 scale, where 1 represents 'Not painful' and 5 represents 'Very painful'. Percentage of participants with each score was reported.
Time Frame: Baseline, Month 6
Population: All enrolled participants. Here 'n' signifies number of participants evaluable at specified time-points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 196
percentage of participants
  Score 1: Baseline (n=196) | 88.8 [83.5 to 92.8]
  Score 1: Month 6 (n=151) | 92.1 [86.5 to 95.8]
  Score 2: Baseline (n=196) | 8.2 [4.7 to 12.9]
  Score 2: Month 6 (n=151) | 6.0 [2.8 to 11.0]
  Score 3: Baseline (n=196) | 1.5 [0.3 to 4.4]
  Score 3: Month 6 (n=151) | 1.3 [0.2 to 4.7]
  Score 4: Baseline (n=196) | 0.5 [0 to 2.8]
  Score 4: Month 6 (n=151) | 0.7 [0 to 3.6]
  Score 5: Baseline (n=196) | 1.0 [0.1 to 3.6]
  Score 5: Month 6 (n=151) | 0 [0 to 0]

20. Secondary Outcome: Percentage of Participants by Injection Site Pain by ESA Type
Description: Assessment was performed by physician via a satisfaction survey on anemia treatment. Participants were asked for the type of ESA received (Mircera, Recormon, Eprex or Aranesp) and to rate their injection site pain on a 1-5 scale, where 1 represents 'Not painful' and 5 represents 'Very painful'. Percentage of participants with each score and ESA type was reported.
Time Frame: Baseline, Month 6
Population: All enrolled participants. Here 'n' signifies number of participants evaluable for specified categories.
Measure: Number; unit: percentage of participants
Arm/Group | Chronic Renal Anemia Participants
Number analyzed (Participants) | 196
percentage of participants
  Mircera: Score 1: Baseline (n=101) | 92.1
  Mircera: Score 2: Baseline (n=101) | 6.9
  Mircera: Score 3: Baseline (n=101) | 1.0
  Mircera: Score 4: Baseline (n=101) | 0
  Mircera: Score 5: Baseline (n=101) | 0
  Mircera: Score 1: Month 6 (n=66) | 97.0
  Mircera: Score 2: Month 6 (n=66) | 3.0
  Mircera: Score 3: Month 6 (n=66) | 0
  Mircera: Score 4: Month 6 (n=66) | 0
  Recormon: Score 1: Baseline (n=34) | 91.2
  Recormon: Score 2: Baseline (n=34 | 5.9
  Recormon: Score 3: Baseline (n=34) | 2.9
  Recormon: Score 4: Baseline (n=34) | 0
  Recormon: Score 5: Baseline (n=34) | 0
  Recormon: Score 1: Month 6 (n=29) | 96.6
  Recormon: Score 2: Month 6 (n=29) | 3.4
  Recormon: Score 3: Month 6 (n=29) | 0
  Recormon: Score 4: Month 6 (n=29) | 0
  Eprex: Score 1: Baseline (n=21) | 71.4
  Eprex: Score 2: Baseline (n=21) | 23.8
  Eprex: Score 3: Baseline (n=21) | 4.8
  Eprex: Score 4: Baseline (n=21) | 0
  Eprex: Score 5: Baseline (n=21) | 0
  Eprex: Score 1: Month 6 (n=19) | 84.2
  Eprex: Score 2: Month 6 (n=19) | 15.8
  Eprex: Score 3: Month 6 (n=19) | 0
  Eprex: Score 4: Month 6 (n=19) | 0
  Aranesp: Score 1: Baseline (n=40) | 87.5
  Aranesp: Score 2: Baseline (n=40) | 5.0
  Aranesp: Score 3: Baseline (n=40) | 0
  Aranesp: Score 4: Baseline (n=40) | 2.5
  Aranesp: Score 5: Baseline (n=40) | 5.0
  Aranesp: Score 1: Month 6 (n=37) | 83.8
  Aranesp: Score 2: Month 6 (n=37) | 8.1
  Aranesp: Score 3: Month 6 (n=37) | 5.4
  Aranesp: Score 4: Month 6 (n=37) | 2.7

ADVERSE EVENTS:
Time Frame: From Baseline up to Month 6
Description: Non-serious adverse events (AEs) were not collected in this study.
Arm/Group | Chronic Renal Anemia Participants
Serious Adverse Events (participants affected / at risk) | 3/196
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chronic Renal Anemia Participants (N=196)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Death (General disorders) | 1

LIMITATIONS AND CAVEATS:
The study was completed as defined in the protocol. Only 196 participants (out of planned 400) were enrolled due to slow recruitment during the study period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.